CLINICAL TRIAL: NCT01798108
Title: A Phase I Open-label, Multicenter, Dose-escalating Study of Radium-223 in Patients With Advanced Skeletal Metastases
Brief Title: Dose Escalation Study of Radium-223 Dichloride in Patients With Advanced Skeletal Metastases
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 15522; ATI-BC-1 (Other: Algeta ASA)
Record Dates: First submitted 2013-01-10; First posted 2013-02-25 (Estimated); Last update posted 2017-05-19 (Actual); Status verified 2017-05

CONDITIONS: Neoplasm Metastasis
Keywords: Advanced skeletal metastases; Radium-223; Radium-223 dichloride; Alpharadin
MeSH Terms: conditions — Neoplasm Metastasis | interventions — radium Ra 223 dichloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Radium-223 dichloride (Experimental): The study had 2 parts. Part 1a was designed with single injections of Radium-223 given to cohorts of 5 patients for each of 5 pre-defined dose levels. Part 1b was designed to retreat and fractionate the dose of Radium-223 in multiple injections.Based on the revised correction factor by calibration, recalculations verified that the single injection doses administered in the part 1a were : 46, 93, 163, 213 and 250 kBq/kg b.w. Two re-treated patients (dose group 6) received a second dose that resulted in a total dose of 250 kBq/kg b.w. The fractionated doses were 1/5 and ½ of the highest dose in part1b (i.e. 250kBq so 5 x 50 and 2 x 125 kBq/kg b.w. respectively).
  Interventions: Radiation: Radium-223 dichloride (BAY88-8223)

INTERVENTIONS:
Radiation: Radium-223 dichloride (BAY88-8223) — - Single injection. Starting dose 46 kBq/kg b.w. Escalating doses 93, 163, 213 and 250 kBq/kg b.w. (9.8.2 Changes in addition to those described in amendments) After completion of the five dose levels above, the protocol was amended and the study extended to include patients to received multiple injections of Radium-223 - Re-treatment: Patients who had earlier been included in the study and received dose levels 46, 93 or 163 kBq/kg b.w. could be given a second injection, provided that the total dose did not exceed 250 kBq/kg b.w. - Fractionated dose (multiple dosing) Patients were given multiple injections in treatment: 5 injections of 50 kBq/kg b.w. at 3 weeks intervals. Patients were given multiple injections in treatment: 2 injections of 125 kBq/kg b.w. at 6 weeks interval

SUMMARY:
A new bone-seeking radiopharmaceutical drug, called Radium-223 dichloride (formerly known as "Alpharadin"), is currently under development. It is an injectable aqueous solution containing radium-223, a radionuclide that emits radiation of another quality and with a different distribution than radiopharmaceuticals currently in use.

After injection of the drug into the blood, a large portion of the drug will accumulate in the bones, and irradiate the skeletal metastases. The drug is expected to be retained longer in the painful sites of bone than in other sites of the body, and may alleviate pain through its radiation. Radium-223 is expected to be both efficacious as regards the targeted localised irradiation, and also to have a favourable safety profile.

The radiopharmaceutical drug Radium-223 has not been given to humans before. In this first clinical study in man, a so-called phase I study, the safety, tolerance and the toxicity of various radioactivity doses of Radium-223 will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 30 years of age
* has histologically or cytologically confirmed breast or prostate carcinoma
* presents with bony metastases, confirmed by scintigraphic imaging within the previous 4 weeks
* relapsing with new foci in the skeleton after previous external radiotherapy
* has a life expectancy of at least 8 weeks (study part Ia), 5 months for study part Ib
* good performance status; ECOG (Eastern Cooperative Oncology Group) status 0-2
* has normal bone marrow, hepatic, renal and cardiac functions
* clinical chemical laboratory values are within pre-specified range, measured within 7 days prior to dosing day
* for female patients: post-menopausal, surgically sterile or taking adequate contraceptive precaution

Exclusion Criteria:

* has previously been included in this study. This criterion is applicable for patients that receive a single injection of the study drug, but not for patients to be re-treated, or for those to receive a fractionated dosing regimen (study part Ib).
* has received an investigational drug in the 4 weeks before or is scheduled to receiving one during or in the 8 weeks after study drug administration. This criterion is applicable for patients that receive a single injection of the study drug and for patients to be re-treated.
* has received any other investigational drug than radium-223 in the 4 weeks before first injection of study drug or is scheduled to receiving one during or in the 8 weeks after the fractionated study drug regimen. This criterion is applicable for patients receiving fractionated dose of the study drug.
* has received chemo-, immuno-, or radiotherapy within the last 4 weeks prior to entry in the study
* has other active, serious, life-threatening disease with a life expectancy of less than 8 weeks
* has any uncontrolled infection
* requires oxygen for pulmonary metastases
* has poor renal function with S-Creatinine >150 mmol/L (males), >100 mmol/L (females)
* has heart insufficiency, Class III or IV NYHA (New York Heart Association)
* is pregnant or lactating
* for female patients: of childbearing potential, and not taking adequate contraceptive measures

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2001-08-14 (Actual); Primary Completion 2003-06-25 (Actual); Study Completion 2003-06-25 (Actual)

PRIMARY OUTCOMES:
Number of participants with predetermined adverse events (dose limiting toxicity [DLT]) as a measure of safety and tolerability while dose escalating | Up to 8 weeks from injection

SECONDARY OUTCOMES:
Blood clearance of radioactivity | 48 hours after the last injection
Quality of Life Questionnaire | 8 weeks after the last injection

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (3):
- Norway (2):
  - The Norwegian Radium Hospital, Oslo
  - University Hospital of North Norway, Tromsø
- Karolinska University Hospital, Stockholm, Sweden

REFERENCES:
- [Background] Nilsson S, Larsen RH, Fossa SD, Balteskard L, Borch KW, Westlin JE, Salberg G, Bruland OS. First clinical experience with alpha-emitting radium-223 in the treatment of skeletal metastases. Clin Cancer Res. 2005 Jun 15;11(12):4451-9. doi: 10.1158/1078-0432.CCR-04-2244. PMID 15958630